CLINICAL TRIAL: NCT03039621
Title: International Multicenter Double-blind Placebo-Controlled Parallel-Group Randomized Clinical Trial of Efficacy and Safety of Ergoferon in the Treatment of Acute Respiratory Viral Infections in Children
Brief Title: Clinical Trial of Efficacy and Safety of Ergoferon in the Treatment of Acute Respiratory Viral Infections in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-ER-009
Record Dates: First submitted 2016-12-28; First posted 2017-02-01 (Estimated); Results first posted 2020-04-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2019-05

CONDITIONS: Acute Respiratory Viral Infections
MeSH Terms: interventions — ergoferon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Ergoferon (Experimental): Tablet for oral use, 1 tablet per intake (outside a meal/feeding). On day 1, five tablets are taken in the first 2 hours (one tablet every 30 min), followed by three more tablets regularly spaced during the rest of the day (total 8 tablets). From day 2, one tablet is taken every 8 hours. The drug is administered outside a meal (in the interval between meals or 15 minutes before meal or fluid intake). Keep the tablet in the mouth, without swallowing, until completely dissolved. For young children (aged 6 months to 3 years old), the tablet is recommended to be dissolved in a small amount (1 tablespoon) of drinking water of room temperature. The therapy lasts for 5 days.
  Interventions: Drug: Ergoferon
- Placebo (Placebo Comparator): Placebo using Ergoferon scheme.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ergoferon — For oral use.
  Arms: Ergoferon
Drug: Placebo — For oral use.
  Arms: Placebo

SUMMARY:
The international multicenter double-blind placebo-controlled randomized clinical study in parallel groups.The objective of this study is to obtain additional data on the efficacy and safety of Ergoferon in the treatment of acute respiratory viral infections (ARVI) in children aged from 6 months to 6 years old.

DETAILED DESCRIPTION:
Study design: international, multicenter double-blind placebo-controlled randomized clinical study in parallel groups.

The study will enroll patients of either gender aged from 6 months to 6 years old with clinical manifestations of ARVI within the first days after the onset of the disease. Patients will be included evenly (1:1 ratio) in accordance with the age group: 6 months - 3 years 11 months 29 days; 4 years - 6 years 11 months 29 days. Signed information sheet for parents/adopters (inform consent form) will be obtained from all participant's parents/ adopters prior to the screening procedures. Medical history, thermometry, patient examination by the doctor, assesment of ARVI symptoms severity and nasopharyngeal swabswill be performed at screening visit (Day 1).

If the inclusion criteria are met and exclusion criteria are absent, the patient is included in the study.

Nasopharyngeal swabs will be analyzed by real-time reverse transcription polymerase chain reaction (RT-PCR) to identify the most common respiratory viruses, including (1) Influenza A virus; (2) Influenza B virus; (3) Influenza A (H1N1)pdm; (4) Human metapneumovirus; (5) Human respiratory syncytial virus; (6) Human rhinovirus; (7) Human adenovirus; (8) Human bocavirus; (9) Human parainfluenza virus 1; (10) Human parainfluenza virus 2; (11) Human parainfluenza virus 3; (12) Human parainfluenza virus 4; (13) Human coronavirus OC43; (14) Human coronavirus 229E; (15) Human coronavirus HKU1; (16) Human coronavirus NL63.

The patients are randomized into one of two groups: the 1st group patients will take Ergoferon according to the dosage regimen for 5 days; the 2nd group patients will take Placebo according to the dosage regimen of Ergoferon for 5 days. Patient's parents/ adoptive parents are provided with diares, where daily in the morning and at hight they record oral temperature (measured by a digital thermometer provided by Sponsor), symptoms of ARVI (according to the 4-points scale), administered drug and concomitant therapy. The doctors instruct parents/ adoptive parents how to fill in the diaries; the first scores of ARVI symptoms severity and oral temperature are made by doctors together with the parents/adoptive parents.

Patients are observed up for 14 days (screening and randomization - up to 1 day, therapy for 5 days, follow-up from 6 to 10 days; delayed telephone "visit" - on day 14).

During the observation period, two visits are planned (at home or at the medical center) on day 3 (Visit 2) and day 6 (Visit 3). If patients still have any symptoms of ARVI/ complications of ARVI, then an additional (unscheduled) Visit 4 is provided on Day 10 of the observation (at the medical center). During Visits 2, 3 (4), doctors carry out an physical examination, record dynamics of ARVI symptoms and concomitant therapy, check patient's diaries, which parents/adoptive parents return back at Visit 3 or 4. At Visit 3 (after 5 days of therapy) compliance with the treatment is additionally assessed. A "telephone visit" (Visit 5, Day 14 ± 1) is carried out to interview parents about the patient's condition, presence/ absence of complications, and possible use of antibiotics.

During the study, symptomatic therapy and therapy for underlying chronic conditions are allowed with the exception of the drugs indicated in the section "Prohibited Concomitant Therapy".

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders aged from 6 months to 6 years old.
2. ARVI based on medical examination: oral temperature of at least 38.0°C at examination + total symptom severity ≥5.
3. The first 24 hours after ARVI onset.
4. Seasonal raise in ARVI incidence.
5. Availability of signed information sheet for parents/adopters(Informed Consent Form) for participation in the clinical trial.

Exclusion Criteria:

1. Suspected pneumonia or bacterial infection (e.g. meningitis, sepsis, otitis media, urinary tract infection, etc.) requiring a prescription of antibacterial product from the first day of the disease.
2. Suspected initial manifestations of diseases with symptoms similar to ARVI at onset (other infectious diseases, flu-like syndrome at the onset of systemic diseases of connective tissue, oncohaematological and other diseases).
3. Clinical symptoms of severe influenza infection/ARVI requiring hospitalization.
4. Medical history of primary and secondary immunodeficiency; oncologic conditions.
5. Aggravation or decompensation of chronic disease (diabetes mellitus, cerebral palsy, cystic fibrosis, primary ciliary dyskinesia, bronchopulmonary dysplasia, malformations of the respiratory and ETN organs/ear, throat, mouth, tongue, larynx, trachea, neck and salivary and thyroid glands, etc.) which affect the patient's ability to participate in the clinical study.
6. Malabsorption syndrome, including congenital or acquired lactase or other disaccharidase deficiency, galactosemia.
7. Allergy/hypersensitivity to any components of the drug product used in the therapy.
8. Course administration of the drug products specified in the section "Prohibited Concomitant Therapy" within two weeks prior to inclusion in the study.
9. Patients whose parents/adoptive parents will not fulfil the requirements during the study or follow the order of administration of the studied drug products from the investigator's point of view.
10. Participation in other clinical trials within 3 months prior to the enrollment in this study.
11. The patient's parent/adoptive parent is a study specialist at the centre and is directly involved in the study or is an immediate family member of the investigator. Spouses parents, children or siblings, regardless of whether they are siblings or adopted are considered immediate family members.
12. The patient's parent/adoptive parent works at OOO "NPF "MATERIA MEDICA HOLDING", i.e. they are employees of the Company, temporary employees on a contract basis or appointed official responsible for conduction of the study or their immediate family members.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 287 (Actual)
Dates: Start 2016-10-07 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-01-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Kazakhstan (3):
  - Kazakh Medical Continuing Education University, Almaty
  - Astana Medical University, Astana
  - Karaganda State Medical University, Karaganda
- Russia (10):
  - Federal State Budgetary Educational Institution of Higher Education "Kazan Medical University" of the Ministry of Healthcare of the Russian Federation, Kazan'
  - Federal State Budgetary Educational Institution of Higher Education "Pirogov Russian National Research Medical University" of the Ministry of Healthcare of the Russian Federation, Moscow
  - Limited Liability Company "Diagnostics and Vaccines", Moscow
  - St. Petersburg State Budgetary Health Care Institution "Сity Polyclinic №44", Moscow
  - Municipal Health Care Institution "City Child Health Clinical Polyclinic №5", Perm
  - State Budgetary Institution of Healthcare of the Samara Region "Samara City Children's Clinical Hospital named after N.N. Willow New, Samara
  - Volgograd State Medical University, Volgograd
  - Yaroslavl State Medical University/Children's Clinic # 5, Yaroslavl
  - Yaroslavl State Medical University/Clinical Hospital # 8, Yaroslavl
  - Municipal autonomous institution "Children's City Clinical Hospital №11", Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Groups:
- Ergoferon: 1 tablet 3 times a day.
  Ergoferon: Inside, orally.
- Placebo: 1 tablet 3 times a day.
  Placebo: Inside, orally.
Period: Overall Study
Arm/Group | Ergoferon | Placebo
Started | 143 | 144
Completed | 131 | 128
Not Completed | 12 | 16
Not completed — Violation of inclusion criteria | 3 | 2
Not completed — Non-compliance with protocol requirement | 4 | 5
Not completed — Necessity to use drugs forbidden by pro | 4 | 7
Not completed — Violation of non-inclusion criteria | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Ergoferon: Ergoferon: Tablet for oral use, 1 tablet per intake (outside a meal/feeding). On day 1, five tablets are taken in the first 2 hours (one tablet every 30 min), followed by three more tablets regularly spaced during the rest of the day (total 8 tablets). From day 2, one tablet is taken every 8 hours.
- Placebo: Placebo: Placebo using Ergoferon scheme.
- Total: Total of all reporting groups
Arm/Group | Ergoferon | Placebo | Total
Number analyzed (Participants) | 143 | 144 | 287
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: ITT sample
  years
    number analyzed (Participants) | 140 | 142 | 282
    (all) | 3.3 (1.7) | 3.4 (1.7) | 3.4 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: ITT sample
  Participants
    number analyzed (Participants) | 140 | 142 | 282
    Female | 73 | 73 | 146
    Male | 67 | 69 | 136
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Kazakhstan | 26 | 25 | 51
  Russia | 117 | 119 | 236

OUTCOME MEASURES:

1. Primary Outcome: Time to Alleviation of All ARVI Symptoms.
Description: Based on patient diary data. Criteria of alleviation of all ARVI symptoms: oral temperature ≤37.5С for 24 hours (without subsequent increase within the observation period) + absence of ARVI symptoms /presence of ARVI symptoms with ≤3-point of the total score (TS) according to the 4-point scale (0 = no symptom; 1 = mild symptom; 2 = moderate symptom; 3 = severe symptom, for each flu-like nonspecific and respiratory symptom). TS ranges from 0 to 30, and the higher scores mean a worse outcome.
Time Frame: 14 days of observation.
Population: ITT sample
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 140 | 142
days | 4.5 [4.2 to 4.8] | 5.2 [4.8 to 5.6]
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Test type: Superiority; p = 0.026, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance equals 0.05

2. Secondary Outcome: Time to Normalization of Body Temperature.
Description: Based on patient diary data. Oral temperature ≤37.5С for 24 hours (without subsequent increase within the observation period).
Time Frame: 14 days of observation.
Population: ITT sample
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 140 | 142
days | 2.8 [2.6 to 3.1] | 3.4 [3.1 to 3.8]
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Test type: Superiority; p = 0.031, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Time to Alleviation of Flu-like Nonspecific Symptoms.
Description: Based on patient diary data. Absence of flu-like nonspecific symptoms/presence of one mild flu-like nonspecific symptom.
Time Frame: 14 days of observation.
Population: ITT sample
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 140 | 142
days | 4.0 [3.7 to 4.3] | 4.7 [4.3 to 5.0]
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Test type: Superiority; p = 0.022, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Time to Alleviation of Respiratory Symptoms.
Description: Based on patient diary data. Absence of respiratory symptoms/presence of one mild respiratory symptom.
Time Frame: 14 days of observation.
Population: ITT sample
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 140 | 142
days | 4.3 [4.0 to 4.6] | 5.0 [4.6 to 5.4]
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Test type: Superiority; p = 0.024, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Flu-like Nonspecific and Respiratory Symptoms Total Score (TS) for Days 2-6.
Description: Based on patient diary data. The total score (TS) ranges from 0 to 30 consisting of 4 flu-like nonspecific (decreased activity/weakness, poor appetite/refusal to eat, sick appearance, sleep disturbance) and 6 respiratory (runny nose, stuffy nose/nasal congestion, sneezing, hoarseness, sore throat, cough) symptoms according to the 4-point scale for each symptom (0 = no symptom; 1 = mild symptom; 2 = moderate symptom; 3 = severe symptom). TS ranges from 0 to 30, and the higher scores mean a worse outcome.
Time Frame: On days 2-6 of the observation period.
Population: ITT sample
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 140 | 142
score on a scale
  Day 2 | 12.0 [11.2 to 12.9] | 13.1 [12.3 to 13.9]
  Day 3 | 8.7 [7.9 to 9.6] | 9.7 [8.8 to 10.6]
  Day 4 | 6.2 [5.4 to 7.0] | 7.1 [6.2 to 7.9]
  Day 5 | 3.9 [3.3 to 4.5] | 5.1 [4.4 to 5.9]
  Day 6 | 2.5 [2.1 to 3.0] | 3.7 [3.1 to 4.4]
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Test type: Superiority; p = 0.0201, Mixed Models Analysis — The p-value associated with "treatment" factor of total severity index of the disease from Day 2 to Day 3, 4, 5 and 6 endpoint between Ergoferon and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction

6. Secondary Outcome: ARVI Severity.
Description: Based on the area under the curve of TS for days 2-6, according to the patient diary. The total score (TS) will be calculated based on the severity of each ARVI symptom (sum of 11 symptoms = body temperature, flu-like nonspecific symptoms (4 symptoms) and respiratory symptoms (6 symptoms) according to the 4-point scale (0 = no symptom; 1 = mild symptom; 2 = moderate symptom; 3 = severe symptom). To calculate TS the absolute oral temperature values, measured in degrees Celsius, will be converted into relative units (or points), given the following gradations: ≤37.5С = 0 point; 37.6-38.1C = 1 point; 38.2-38.8C = 2 points; ≥38.90С = 3 points. For total score minimum and maximum scores are 0 and 33, where higher values represent a worse outcome.
Time Frame: On days 2-6 of the observation period.
Population: ITT sample
Measure: Mean (95% Confidence Interval); unit: score on a scale*day
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 140 | 142
score on a scale*day | 39.6 [36.4 to 42.8] | 44.6 [41.2 to 48.1]
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Test type: Superiority; p = 0.046, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Percentage of Recovered Patients.
Description: Based on patient diary data. Criteria of recovery/alleviation of all ARVI symptoms: oral temperature ≤37.5С for 24 hours (without subsequent increase within the observation period) + absence of ARVI symptoms /presence of ARVI symptoms with ≤3-point of the total score (TS) according to the 4-point scale for each flu-like nonspecific and respiratory symptom (0 = no symptom; 1 = mild symptom; 2 = moderate symptom; 3 = severe symptom, for each flu-like nonspecific and respiratory symptom).
Time Frame: On days 2-6 of the observation period.
Population: ITT sample
Measure: Count of Participants; unit: Participants
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 140 | 142
Participants
  Day 2 | 20 | 20
  Day 3 | 37 | 35
  Day 4 | 72 | 61
  Day 5 | 102 | 91
  Day 6 | 119 | 98
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Test type: Superiority; p = 0.0025, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Ergoferon vs Placebo; Test type: Other — Test for assessing the homogeneity of the odds ratio in several 2 × 2 contingency tables; p = 0.22, Breslow-Day test

8. Secondary Outcome: Rates of Antipyretics Use Per Patient.
Description: Based on patient diary data. The number of intakes of prescribed antipyretics.
Time Frame: On days 1- 5 of the treatment period.
Population: ITT sample
Measure: Mean (95% Confidence Interval); unit: number per patient
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 140 | 142
number per patient
  Day 1 | 1.5 [1.3 to 1.6] | 1.6 [1.4 to 1.7]
  Day 2 | 1.0 [0.9 to 1.2] | 1.2 [1.0 to 1.4]
  Day 3 | 0.4 [0.2 to 0.5] | 0.5 [0.4 to 0.6]
  Day 4 | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.3]
  Day 5 | 0.0 [0.0 to 0.1] | 0.1 [0.0 to 0.2]
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Test type: Superiority; p = 0.0037, Mixed Models Analysis — The p-value associated with "treatment" factor of total severity index of the disease from Day 1 to Day 2, 3 and 4 endpoint between Ergoferon and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction

9. Secondary Outcome: Percentage of Patients With Worsening of Illness.
Description: Based on patient diary data. The disease worsening: ARVI complications, including those requiring antibiotics; hospitalization).
Time Frame: 14 days of observation peiod.
Population: ITT sample
Measure: Count of Participants; unit: Participants
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 140 | 142
Participants | 1 | 19
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Test type: Superiority; p = 0.0001, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse/Serious adverse events were registered during 14 days (during the treatment and follow-up periods).
Description: Adverse/Serious adverse events were registered in patients of the Safety population (n=287).
Arm/Group | Ergoferon | Placebo
All-Cause Mortality (participants affected / at risk) | 10/143 | 27/144
Serious Adverse Events (participants affected / at risk) | 0/143 | 0/144
Other Adverse Events (participants affected / at risk) | 10/143 | 27/144
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ergoferon (N=143) | Placebo (N=144)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Bilateral cervical lymphadenitis
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) — Tachycardia NOS
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) — Eyelid oedema
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (2) — Diarrhoea
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) — Vomiting
Teething (Gastrointestinal disorders) | 0 (0) | 1 (1) — Teething syndrome
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Abdominal pain
Hyperthermia (General disorders) | 0 (0) | 1 (1) — Hyperthermia sudden
Condition worsened (General disorders) | 1 (1) | 3 (3) — Condition worsened
Adenoiditis (Infections and infestations) | 1 (1) | 8 (8) — Adenoiditis
Bronchitis (Infections and infestations) | 0 (0) | 4 (4) — Obstructive bronchitis
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) — Acute gastroenteritis
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) — Acute laryngotracheitis
Otitis media acute (Infections and infestations) | 0 (0) | 2 (2) — Acute mucoid otitis media
Otitis media acute (Infections and infestations) | 1 (1) | 2 (2) — Otitis media acute
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) — Acute rhinitis
Adenoviral upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) — Adenoviral upper respiratory infection
Gastroenterocolitis (Infections and infestations) | 0 (0) | 1 (1) — Gastroenterocolitis
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) — Herpes labialis
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0) — Infectious mononucleosis
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 2 (2) — Pharyngotonsillitis
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Post procedural vomiting
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Myalgia
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Muscle twitching
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Acute torticollis
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Nasal discharge
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Cough aggravated
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Dermatitis atopic aggravated
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Urticaria
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash desquamating
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Localised rash

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT03039621/Prot_SAP_000.pdf